CLINICAL TRIAL: NCT04844580
Title: A Comparative, Multicenter, Placebo-Controlled, Double-Blind Phase II Clinical Trial Evaluating the Efficacy, Safety and Tolerability of Inhaled Aviptadil in Patients 18 Years and Older With COVID-19 Pulmonary Involvement - HOPE
Brief Title: A Clinical Study Evaluating Inhaled Aviptadil on COVID-19
Acronym: HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centurion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-AY001-HOPE
Record Dates: First submitted 2021-03-25; First posted 2021-04-14 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Aviptadil; Inhaled; COVID-19; Pandemic
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: In the study, patients will be randomized in a ratio of 1: 1 into two arms, standard medical therapy + placebo versus standard medical therapy + inhaled Aviptadil arms. Randomization will be carried out by the block randomization method.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment + Placebo (Placebo Comparator): Standard medical treatment, as deemed appropriate by physicians, is going to be according to the Turkish Republic COVID-19 (SARS-CoV-2 INFECTION) ADULT PATIENT TREATMENT GUIDELINES published by the Ministry of Health, General Directorate of Public Health. The management of all additional complications and / or symptoms that develop in patients will be managed in the same way as specified in these guidelines. If these guidelines are changed by the Turkish Republic Ministry of Health General Directorate of Public Health, a protocol amendment will be planned. The necessary changes within the scope of urgent security measures will be reflected in the standard treatment in accordance with the necessary regulations.
  Interventions: Drug: Placebo
- Standard Treatment + Inhaled Aviptadil (Experimental): In addition to the standard medical treatment mentioned above, patients randomized to this arm will be given Inhaled Aviptadil 2 times a day, 30 minutes apart. Aviptadil treatment is aimed to be a minimum of 7 days and a maximum of 14 days. Aviptadil will be discontinued in patients who do not heal after 14 days. The dose of inhaled Aviptadil was determined by evaluating the results of the Phase 1 and Phase 2 studies.
  Interventions: Drug: Inhaled Aviptadil

INTERVENTIONS:
Drug: Inhaled Aviptadil — Aviptadil is the synthetic analogue of the Vasoactive Intestinal Peptide (VIP), a biologically active 28 amino acid natural peptide that is endogenously synthesized in humans. It is one of the signaling molecules of the neuroendocrine immune network and has vasodilator, anti-proliferative, anti-inflammatory and immunomodulatory properties.
  Arms: Standard Treatment + Inhaled Aviptadil
Drug: Placebo — Aviptadil Placebo will be used for this arm.
  Arms: Standard Treatment + Placebo

SUMMARY:
This study is a multicenter, prospective, placebo-controlled, comparative, randomized, double-blind local phase II clinical trial. Duration of study is 18 months. In the study, patients will be randomized in a ratio of 1: 1 into two arms, standard medical therapy + placebo versus standard medical therapy + inhaled Aviptadil arms. Randomization will be carried out by the block randomization method. In the event that patients need intensive care in the study, the patients will be taken into intensive care unit and excluded from the study and their treatment will be continued in the intensive care unit as deemed appropriate by the physician and it is foreseen that inhaled Aviptadil will be used for a period of minimum 7 and maximum 14 days. Aviptadil will be discontinued in patients who do not heal after 14 days. This study includes 8 visits, consisting of a total of 7 physical visits and 1 phone follow-up visit. The study period will be 6 months for each patient. Patient recruitment is planned to take 12 months. Study centers will be asked to use investigational products for their patients who sign the informed consent form for 12 months. The study population will consist of patients 18 years of age and older with COVID-19 pulmonary involvement and hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

1.18 years and older women or men, under 70 years old

2.Patients with positive SARS-CoV-2 real time PCR result and an appearance in line with COVID-19 pneumonia on thorax CT

3. Need for oxygen support or SpO2 <94 in room air

4. Patients who can use a nebulizer (with assistance when necessary)

5.Patients who are willing and capable (mentally and physically) who can sign a written informed consent form, to participate in all aspects of the study, to participate in the planned visits and to comply with the terms of the protocol.

Exclusion Criteria:

1. Intensive care admission
2. The need for mechanical ventilation
3. Patients with previously known organ (kidney, heart and liver) failure

   * To be determined as previously known heart failure (EF <30), previously known liver failure (Child-Pugh C) and previously known renal failure (Cr.clerance <30).
4. COVID-19 disease with no indication for hospitalization
5. Participants in another clinical trial
6. Pregnancy or lactation
7. Solid organ or stem cell transplantation story
8. Patients with collagen tissue disease
9. Use of immunosuppressive therapy
10. Procalcitonin ≥2 (baseline visit)
11. Under 18 years old
12. Those who had myocardial infarction in the last 3 months
13. Those who do not have the capacity to understand the possible results, scope and nature of the study due to legal insufficiency and / or other reasons.
14. Those who, in the opinion of the investigator, cannot continue the treatment protocol regularly or cannot cooperate
15. Presence of malignancy
16. Patients with neurological diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 6 months
  Being discharged within 30 days of starting treatment, no need for oxygen support

SECONDARY OUTCOMES:
Time to discharge of patients | 6 months
The rate of patients entering intensive care | 6 months
Patients' rate of needing mechanical ventilation | 6 months
Change in SpO2 (measured by pulse oximetry) | 6 months
Normalization in body temperature | 14 days
Dyspnea Scale (Modified Borg Dyspnea Scale (MBS) | 6 months
6-minute walking test | 28 days
The time it takes for patients to improvement of their symptoms (cough, shortness of breath) | 6 months
The time it takes for the PCR to become negative | 14 days
Sequelae and recovery rates in control thorax computed tomography at the end of month 1 and 6 months | 6 months
Need for re-hospitalization | 6 months
Normalization in laboratory results of blood parameters (PT, aPTT, D-dimer, Ferritin, Lymphocyte Count, CRP) | 28 days
Normalization in laboratory results of biochemistry parameters (Glucose, ALT, AST, LDH, Total Bilirubin, Total Protein, Albumin, Alkaline Phosphatase, GGT, Sodium, Potassium, Calcium, Phosphor, CPK, Magnesium, eGFR, BUN, Uric Acid, Creatinine Clearance) | 28 days
Mortality rate | 6 months
Normalization in Blood Pressure | 14 days
Normalization in Respiration Rate/Minute | 14 days
Normalization in SpO2 | 14 days

CONTACTS AND LOCATIONS:
Locations (9):
- Turkey (Türkiye) (9):
  - Başkent University School of Medicine, Ankara
  - Hacettepe University School of Medicine, Ankara
  - Dicle Üniversitesi Tıp Fakültesi Hastanesi, Diyarbakır
  - Başakşehir Çam ve Sakura Şehir Hastanesi, Istanbul
  - Health Sciences University Yedikule Training and Research Hospital, Istanbul
  - Prof. Dr. Feriha Öz Acil Durum Hastanesi, Istanbul
  - Prof. Dr. Murat Dilmener Acil Durum Hastanesi, Istanbul
  - Kocaeli Üniversitesi Tıp Fakültesi Hastanesi, Kocaeli
  - Karadeniz Teknik Üniversitesi Tıp Fakültesi Hastanesi, Trabzon

IPD SHARING:
Plan to Share IPD: No